CLINICAL TRIAL: NCT06757322
Title: Comparison of Single Needle-Double Cannula and Double Needle Arthrocentesis in Temporomandibular Joint Disorders
Brief Title: Comparing Single Needle and Double Needle Arthrocentesis for Temporomandibular Joint Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YYU/06/04.03.2020
Record Dates: First submitted 2024-12-18; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: TMJ Disc Disorder
Keywords: arthrocentesis; disc displacement without reduction; temporomandibular joint disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-needle double cannula arthrocentesis group (Active Comparator): In the single-needle group, two needles were bent (from their lower parts) before the procedure and their pointed ends were joined by placing acrylic on the plastic parts from a single point. The resulting combined needle was directed to the upper joint space and washed.
  Interventions: Procedure: Singel Needle Double Cannula TMJ Arthrocentesis
- Double-needle arthrocentesis group (Active Comparator): Two needles were inserted into the TMJ and washed.
  Interventions: Procedure: Double Needle TMJ Arthrocentesis

INTERVENTIONS:
Procedure: Singel Needle Double Cannula TMJ Arthrocentesis — Artocentesis describes the lavage of the TMJ by introducing a saline/ringer lactate solution through a needle inserted into the upper joint cavity. TMJ arthrocentesis was first introduced as a double needle entry method by Nitzan et al in 1991. The single needle technique was developed by Singh and Varghese and introduced in 2013. The single needle method is a more simplified modification of the first method.
  Arms: single-needle double cannula arthrocentesis group
Procedure: Double Needle TMJ Arthrocentesis — Artocentesis describes the lavage of the TMJ by introducing a saline/ringer lactate solution through a needle inserted into the upper joint cavity. TMJ arthrocentesis was first introduced as a double needle entry method by Nitzan et al in 1991.
  Arms: Double-needle arthrocentesis group

SUMMARY:
The purpose of this study was to compare the clinical success and efficacy of single-needle, double-cannula arthrocentesis with conventional arthrocentesis techniques in patients with temporomandibular joint disorders. Patients with nonreducible disc displacement complained of limited mouth opening and/or pain. All treated patients had baseline and follow-up (with mouth opening and VAS). Comparisons were made within and between groups.

DETAILED DESCRIPTION:
The patients included in the study were evaluated in the preoperative, 1week, 1-3, and 6 months after the procedure. Double-needle group: two needles were inserted into the joint and washed. In the single-needle group, two needles were bent (from their lower parts) before the procedure and their pointed ends were joined by placing acrylic on the plastic parts from a single point. The resulting combined needle was directed to the upper joint space and washed. 13 underwent single-needle double cannula arthrocentesis and 15 underwent double needle arthrocentesis.

ELIGIBILITY:
Inclusion Criteria:

* with complaints of pain and restricted mouth opening and who had not received any previous treatment.
* Patients with a diagnosis of disc displacement without reduction characterized by persistent or frequent TMJ pain, history of joint clicking, limited mouth opening with deviation to the affected side, limited lateral movement to the opposite side, limited protrusive movements with deviation to the affected side were included.

Exclusion Criteria:

* Patients with systemic inflammatory joint disease, facial growth disorder, and direct trauma to the TMJ were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
change in mouth opening | Until the 6th month after TMJ Arthrocentesis
  The maximum mouth opening of the patients was noted in centimeters before arthrocentesis and in the control sessions, and the changes between the sessions were compared.
VAS Pain Scor | Until the 6th month after TMJ Arthrocentesis
  The VAS pain assessments of the patients before and during the arthrocentesis and control sessions were noted and changes between sessions were compared. The VAS score is an assessment in which we note the patient's pain assessment between 0 and 10. '0' means no pain, while '10' means the worst possible pain. As the number increases, it indicates that the patient's pain increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl Üniversitesi Diş Hekimliği Fakültesi, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senturk MF, Cambazoglu M. A new classification for temporomandibular joint arthrocentesis techniques. Int J Oral Maxillofac Surg. 2015 Mar;44(3):417-8. doi: 10.1016/j.ijom.2014.11.014. Epub 2014 Dec 17. No abstract available. PMID 25529932
- [Background] Sequeira J, Rao BHS, Kedia PR. Efficacy of Sodium Hyaluronate for Temporomandibular Joint Disorder by Single-Puncture Arthrocentesis. J Maxillofac Oral Surg. 2019 Mar;18(1):88-92. doi: 10.1007/s12663-018-1093-4. Epub 2018 Feb 27. PMID 30728698
- [Background] Nagori SA, Jose A, Roychoudhury A. Comparison of intraoperative outcomes with single and double puncture techniques of arthrocentesis of the temporomandibular joint. Br J Oral Maxillofac Surg. 2020 Oct;58(8):928-932. doi: 10.1016/j.bjoms.2020.04.011. Epub 2020 Jul 16. PMID 32684314
- [Background] Folle FS, Poluha RL, Setogutti ET, Grossmann E. Double puncture versus single puncture arthrocentesis for the management of unilateral temporomandibular joint disc displacement without reduction: A randomized controlled trial. J Craniomaxillofac Surg. 2018 Dec;46(12):2003-2007. doi: 10.1016/j.jcms.2018.10.015. Epub 2018 Oct 26. PMID 30446325
- [Background] Nagori SA, Bansal A, Jose A, Roychoudhury A. Comparison of outcomes with the single-puncture and double-puncture techniques of arthrocentesis of the temporomandibular joint: An updated systematic review and meta-analysis. J Oral Rehabil. 2021 Sep;48(9):1056-1065. doi: 10.1111/joor.13228. Epub 2021 Jul 23. PMID 34273184
- [Background] Senturk MF, Tuzuner-Oncul AM, Cambazoglu M. Prospective short term comparison of outcomes after single or double puncture arthrocentesis of the temporomandibular joint. Br J Oral Maxillofac Surg. 2016 Jan;54(1):26-9. doi: 10.1016/j.bjoms.2015.11.004. Epub 2015 Nov 30. PMID 26782027
- [Background] Bayramoglu Z, Tozoglu S. Comparison of single- and double-puncture arthrocentesis for the treatment of temporomandibular joint disorders: A six-month, prospective study. Cranio. 2021 Mar;39(2):151-156. doi: 10.1080/08869634.2019.1603796. Epub 2019 Apr 25. PMID 31021311
- [Background] Talaat W, Ghoneim MM, Elsholkamy M. Single-needle arthrocentesis (Shepard cannula) vs. double-needle arthrocentesis for treating disc displacement without reduction. Cranio. 2016 Sep;34(5):296-302. doi: 10.1080/08869634.2015.1106810. Epub 2016 Apr 13. PMID 27077267
- [Background] Senturk MF, Yazici T, Gulsen U. Techniques and modifications for TMJ arthrocentesis: A literature review. Cranio. 2018 Sep;36(5):332-340. doi: 10.1080/08869634.2017.1340226. Epub 2017 Jun 15. PMID 28618972
- [Background] Siewert-Gutowska M, Pokrowiecki R, Kaminski A, Zawadzki P, Stopa Z. State of the Art in Temporomandibular Joint Arthrocentesis-A Systematic Review. J Clin Med. 2023 Jun 30;12(13):4439. doi: 10.3390/jcm12134439. PMID 37445474
- [Background] Alkan A, Bas B. The use of double-needle canula method for temporomandibular joint arthrocentesis: clinical report. Eur J Dent. 2007 Jul;1(3):179-82. PMID 19212563
- [Background] Tvrdy P, Heinz P, Pink R. Arthrocentesis of the temporomandibular joint: a review. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2015 Mar;159(1):31-4. doi: 10.5507/bp.2013.026. Epub 2013 Apr 10. PMID 23579112

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT06757322/Prot_SAP_000.pdf